CLINICAL TRIAL: NCT01927926
Title: The Effects of Consuming Between- Meal, High Protein Polydextrose Containing Snack Bars on Subjective Satiety, Energy Intake and Metabolic Responses.
Brief Title: The Effects of Consuming Whey Protein Polydextrose Snacks on Appetite and Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Mars, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: A/5/2008
Record Dates: First submitted 2013-08-14; First posted 2013-08-23 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Obesity
Keywords: Energy intake; appetite; satiety; gut hormones
MeSH Terms: conditions — Obesity | interventions — Whey

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whey-protein & polydextrose snack (Experimental): Whey-protein & polydextrose snack bar.
  Interventions: Dietary Supplement: Whey-protein & polydextrose snack
- Control snack (Placebo Comparator): Control snack bar containing minimal protein and not polydextrose.
  Interventions: Dietary Supplement: Control snack

INTERVENTIONS:
Dietary Supplement: Whey-protein & polydextrose snack — Subjects will consume one snack bar as a between-meal mid-morning snack daily for 15 days.
  Arms: Whey-protein & polydextrose snack
Dietary Supplement: Control snack — Subjects will consume one snack bar as a between-meal mid-morning snack daily for 15 days.
  Arms: Control snack

SUMMARY:
Developing functional foods that enhance satiety may be beneficial to individuals to help manage body weight.

We have previously shown that consuming a mid-morning liquid preload with increasing proportion of energy derived from whey protein and addition of polydextrose reduced voluntary energy intake at a lunchtime meal compared to a liquid preload of the same energy content but lower in protein and containing no polydextrose.

This study aims to investigate if these results can be replicated when the preload is in the form of a snack bar. We will also investigate whether the daily consumption of the snack bar has an effect on energy intake, subjective appetite and metabolic parameters compared to a control snack of the same energy but with a minimal protein content and without the addition of polydextrose.

We hypothesize that the whey protein polydextrose snack will reduce voluntary energy intake at a subsequent test meal, suppress subjective appetite ratings compared with the control snack bar.

DETAILED DESCRIPTION:
Background:

Developing functional food products that enhance satiety, suppress appetite, and reduce subsequent voluntary food intake to a greater extent than a similar energy matched food product, may be useful to help consumers adhere to energy restricted diets and optimize successful body weight management. A range of foods and food constituents have been reported to have the potential to produce short term changes in appetite and energy intake. However, the effects of consuming foods containing such ingredients on appetite, energy intake over the longer term is unclear.

We have previously shown that consuming a mid-morning liquid preload with increasing proportion of energy derived from whey protein and addition of polydextrose reduced voluntary energy intake at a lunchtime meal compared to a liquid preload of the same energy content but lower in protein and containing no polydextrose.

Aims:

This study aims to investigate if previous findings can be replicated using solid snack bars containing whey protein and polydextrose. We will also investigate whether the daily consumption of the snack bar has an effect on energy intake, subjective appetite and metabolic and endocrine responses.

Methods:

Using a double blind, randomized cross-over design, 10 healthy lean male subjects will consume a whey protein-polydextrose bar and an iso-energetic control bar as a mid-morning, between-meal snack for 14 consecutive days. The two intervention phases will be separated by a 2-wk washout period. On the first (day 1) and the last day (day 15) of each intervention phase, subjective appetite, voluntary food intake, blood metabolite and endocrine responses to the snacks will be assessed under laboratory conditions. Additionally, participants will be asked to record free-living food intake on days 4, 8 and 12 of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-25 kg/m2

Exclusion Criteria:

* Smokers
* BMI <18 > 25 kg/m2
* Dieting or weight loss
* Presence of disease (e.g. diabetes, cardiovascular disease, cancer etc)
* Currently regularly taking medications
* Restrained eaters (defined as restraint score >7 on TFEQ)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-05; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Energy intake at an ad libitum lunchtime test meal | Day 1
  Energy intake at a lunchtime test meal served 90 min following the consumption of the snack bar on day 1.

SECONDARY OUTCOMES:
Energy intake at an ad libitum lunchtime test meal | Day 15
  Energy intake at a lunchtime test meal served 90 min following the consumption of the snack bar on day 15.
Subjective appetite responses | Day 1
  Subjective appetite ratings (hunger, fullness, desire to eat, thirst and nausea) will be recorded when subjects arrive at the laboratory (fasting), prior to the consumption of the snack (-15min), immediately following the consumption of the snack (0 min) and at 30, 60 and 90 min later on day 1.
Remainder of the day energy intake | Day 1
  Subjects will record all foods and drinks consumed after they leave the laboratory, for the remainder of the day on day 1 in a food diary provided.
  Total daily energy intake will be calculated from the sum of energy from foods consumed in the laboratory and foods and drinks recorded in the diary.
Free living energy intake | Day 4
  Subjects will record all foods and drinks consumed on day 4 of the free-living phase of the intervention in a food diary provided.
Free living energy intake | Day 8
  Subjects will record all foods and drinks consumed on day 8 of the free-living phase of the intervention in a food diary provided.
Free living energy intake | Day 12
  Subjects will record all foods and drinks consumed on day 12 of the free-living phase of the intervention in a food diary provided.
Subjective appetite responses | Day 15
  Subjective appetite ratings (hunger, fullness, desire to eat, thirst and nausea) will be recorded when subjects arrive at the laboratory (fasting), prior to the consumption of the snack (-15min), immediately following the consumption of the snack (0 min) and at 30, 60 and 90 min later on day 15.
Remainder of the day energy intake | Day 15
  Subjects will record all foods and drinks consumed after they leave the laboratory, for the remainder of the day on day 15 in a food diary provided.
  Total daily energy intake will be calculated from the sum of energy from foods consumed in the laboratory and foods and drinks recorded in the diary.

OTHER OUTCOMES:
Metabolic responses | Day 1
  Blood samples will be collected in response to the snack bars on day 1 and analyzed for glucose, insulin and ffa.
Metabolic responses | Day 15
  Blood samples will be collected in response to the snack bars on day 15 and analyzed for glucose, insulin and ffa.
Endocrine responses | Day 1
  Blood samples will be collected in response to the snack bars on day 1 and analyzed for GLP-1, PYY and ghrelin.
Endocrine responses | Day 15
  Blood samples will be collected in response to the snack bars on day 15 and analyzed for GLP-1, PYY and ghrelin.

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Macdonald, Phd, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

REFERENCES:
- [Derived] Astbury NM, Taylor MA, French SJ, Macdonald IA. Snacks containing whey protein and polydextrose induce a sustained reduction in daily energy intake over 2 wk under free-living conditions. Am J Clin Nutr. 2014 May;99(5):1131-40. doi: 10.3945/ajcn.113.075978. Epub 2014 Mar 26. PMID 24670946